CLINICAL TRIAL: NCT06381908
Title: The Effects of Combined Energy and Carbohydrate Restriction on Exercise Capacity and Health in Overweight Women
Brief Title: The Effects of Combined Energy and Carbohydrate Restriction on Exercise Capacity
Acronym: CHO-EX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Southern Denmark (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-19-24
Record Dates: First submitted 2024-04-05; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Overweight and Obesity
Keywords: Physical activity; Metabolism; Physical capacity; Macronutrients; Carbohydrate; Diet
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study is performed as a randomized single-blinded parallel group design. Randomization is performed into two groups using minimization based on a predetermined estimated VO2max middle value of 30.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is labelled as a single-blinded study because the investigators are blinded to the group allocation (the group allocation and diet handling is managed by a researcher not involved in other aspects of the data collection or processing). The participants are not informed about their allocated condition, however, it is conceivably possible for them to recognize this based on the food provided. However, the direction of the hypothesis will not be evident to the participants. Moreover, we include questionnaires before the post-tests related to their perceived diet allocation and their perception of the effect of the diet on the test assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-carbohydrate calorie-restriction (Active Comparator): Minimum of 3 g carbohydrate/kg body weight/day and a ~1000 kcal calorie restriction
  Interventions: Other: Calorie-restriction with low carbohydrate
- Moderate-carbohydrate calorie-restriction (Experimental): Maximum of 1 g carbohydrate/kg body weight/day and a ~1000 kcal calorie restriction
  Interventions: Other: Calorie-restriction with moderate carbohydrate

INTERVENTIONS:
Other: Calorie-restriction with low carbohydrate — Calorie-restriction and low carbohydrate availability
  Arms: Low-carbohydrate calorie-restriction
Other: Calorie-restriction with moderate carbohydrate — Calorie-restriction and moderate carbohydrate availability
  Arms: Moderate-carbohydrate calorie-restriction

SUMMARY:
The effect of calorie restriction combined with low or moderate carbohydrate availability on exercise capacity, metabolism and metabolic health indicators will be measured in a randomized parallel group design. Forty overweight (BMI 25-30) and relatively inactive women (20-35 of age) will be included. These will be randomized into one of two experimental groups both receiving a calorie-restricted diet (-1000 kcal) combined with either low carbohydrate availability or moderate carbohydrate availability across a 10 day period. Laboratory-based physical capacity tests and blood and muscle sampling will be performed before and after the intervention. In addition, an additional follow-up test day will be performed after continuing the diet for another 48 h and then standardizing the pre-testing carbohydrate availability before repeating the tests of physical capacity.

DETAILED DESCRIPTION:
Overweight (BMI 25-30), but healthy premenopausal women aged 20-35 years (n=40) will be included in the trial, which is structured as a randomized, parallel group design where participants are randomized to either consume a hypocaloric diet (-1000 kcal) with concurrent carbohydrate restriction (low carbohydrate, L-CHO, n=20) or a similar hypocaloric diet with moderate carbohydrate availability (moderate carbohydrate, M-CHO, n=20). The trial will be single-blinded since it might be transparent to the participants which diet they are consuming, whereas the test personnel collecting and processing test results will be blinded to diet allocation. Diet handling will be managed by specific individuals in the research group who do not partake in executing the physical capacity tests. Additionally, the direction of the trial's primary hypothesis will not be disclosed to the participants to avoid creating preconceived expectations about the effects.

After an initial screening interview and two familiarization visits, participants will complete the intervention period consisting of 10 days with the allocated diet manipulation with preceding and subsequent test days with a series of tests. The tests before and after each test period include measurements of the participants' physical capacity level and energy metabolism in the laboratory as well as blood and muscle sampling. In addition, resting metabolism and body composition will be measured. During each test period, participants' habitual activity level will be monitored with an accelerometer attached to the wrist (Axivity). There will also be monitoring of the activity level with an accelerometer in a 7-day cycle before the start of the trial as a baseline measurement.

Similarly, a glucose monitor will be placed on the upper arm for continuous glucose readings via a Freestyle Libre2 sensor during the trial period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-35
* BMI: 25-30

Exclusion Criteria:

* Irregular menstruation within the last 6 months (shorter end 24 days or longer end 35 days cycle)
* Injuries / pain in the lower body, which prevents participation in intense cycling
* Medication consumption that may affect primary outcome measures.
* Smoking
* Pregnancy
* Systematic physical activity more than 2 hours per week

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Time to exhaustion | Pre, post (day 11 of the intervention) and follow-up (day 2 after the post measurement)
  Time to exhaustion at 85% VO2max
Sprint performance | Pre, post (day 11 of the intervention) and follow-up (day 2 after the post measurement)
  Peak and mean 15-s sprint performance
Exercise tolerance | Pre, post (day 11 of the intervention) and follow-up (day 2 after the post measurement)
  Ratings of perceived exertion (Borg scale) during standardized-intensity exercise from 6 (lowest exertion) to 20 (highest exertion)
Muscle glycogen levels | Pre and post (day 11 of the intervention)
  Muscle glycogen levels obtained from biopsy sample

SECONDARY OUTCOMES:
Physical activity level | During the intervention (days 1 to 11 of the intervention)
  Measured with accelerometer during the intervention
Maximal fat oxidation capacity | Pre, post (day 11 of the intervention) and follow-up (day 2 after the post measurement)
  Maximal fat oxidation measured in the laboratory
Muscle metabolic enzyme activity | Pre and post (day 11 of the intervention)
  Activity of key enzymes involved in carbohydrate and fat metabolism
Blood lipid profile | Pre and post (day 11 of the intervention)
  High-density lipoproteins, low-density lipoproteins, very-low-density lipoproteins, cholesterol, free fatty acids and triglycerides
Continuous glucose levels | 14 days from the day before the intervention, throughout the intervention (days 1 to 11) and 2 days after the intervention (follow-up)
  Glucose levels measured continuously across the trial + during exercise tests
Fasting blood glucose and insulin | Pre and post (day 11 of the intervention)
  Insulin sensitivity (Homa 2 IR)
Long-term glycemic control (HbAc1) | Pre and post (day 11 of the intervention)
  Measured from fasting blood

CONTACTS AND LOCATIONS:
Locations (1):
- Section for Sport Science, Department of Public Health, Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided